CLINICAL TRIAL: NCT01827761
Title: Assessment of the Effectiveness of Chemotherapy Teaching: BrUOG 258
Status: Completed | Type: Observational
Sponsor: Brown University (Other)
Collaborators: Rhode Island Hospital (Other); The Miriam Hospital (Other); Fatima Memorial Hospital (Other); Roger Williams Medical Center (Other); Lifespan (Other)
Responsible Party: Sponsor
Other Study IDs: 258
Record Dates: First submitted 2013-04-04; First posted 2013-04-10 (Estimated); Last update posted 2022-02-24 (Actual); Status verified 2022-02

CONDITIONS: Cancer
Keywords: chemotherapy teaching; questionnaire
MeSH Terms: conditions — Neoplasms | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Questionnaire: After informed consent for this study is obtained, patients will be given questionnaire #1 that includes rating their knowledge of the side effects of treatment, their understanding of the treatment schedule, what do in the event of complication, how to reach the medical team and an assessment of the level of anxiety. The questionnaire will be repeated at day 1 of the first chemotherapy treatment to assess the effectiveness of the teaching session. In addition, questionnaire #3 will be administered at day 1 of cycle 2 of their first chemotherapy.
  Interventions: Behavioral: Questionnaire

INTERVENTIONS:
Behavioral: Questionnaire — After informed consent for this study is obtained, patients will be given questionnaire #1 that includes rating their knowledge of the side effects of treatment, their understanding of the treatment schedule, what do in the event of complication, how to reach the medical team and an assessment of the level of anxiety. The questionnaire will be repeated at day 1 of the first chemotherapy treatment to assess the effectiveness of the teaching session. In addition, questionnaire #3 will be administered at day 1 of cycle 2 of their first chemotherapy.

SUMMARY:
This study will evaluate whether chemotherapy teaching sessions improves patient's knowledge, preparedness and anxiety in relation to chemotherapy. This study will also evaluate the effect of age, race, native language, education level, type of cancer and chemotherapy regimen on the oncology teaching session.

DETAILED DESCRIPTION:
Chemotherapy teaching sessions, often coordinated in the outpatient setting by nursing personnel, are meant to educate patients about the chemotherapy they will be receiving. Education topics include an understanding of side effects, treatment schedule, medications to treat side effects and how to contact the oncology team if adverse events develop. Some of these issues are addressed in the American Society of Clinical Oncology's Quality Oncology Practice Initiative (QOPI). This study will perform an analysis of the teaching process that is provided prior to chemotherapy administration.

This study will provide data for each participating hospital to individually assess their teaching process. Multivariate analysis can be performed to evaluate whether age, sex, native, language, race highest level of education, cancer type, chemotherapy regimen, institution where chemotherapy will be administered, and type of personnel performing the teaching visit, influences the effectiveness of the teaching visit. In addition, results can be compared across different hospitals.This analysis may lead to improvements in each hospital's chemotherapy teaching practices and lead to advances in patient's cognitive and emotional preparedness.

ELIGIBILITY:
Inclusion Criteria:

* Patients > 18 years of age who will be receiving chemotherapy (including targeted anticancer therapy) at a Brown University Oncology Research Group Affiliated Hospital for a period of 1-year after study activation.
* Patients who will be undergoing a chemotherapy teaching session at an institution affiliated with the Brown University Oncology Research Group.
* No prior chemotherapy or targeted anticancer treatment.
* Signed informed consent

Exclusion Criteria:

Patients must meet eligibility criteria

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Cancer Clinics
Sampling Method: Non-Probability Sample
Enrollment: 196 (Actual)
Dates: Start 2011-10; Primary Completion 2014-05 (Actual); Study Completion 2014-05 (Actual)

PRIMARY OUTCOMES:
Evaluate whether chemotherapy teaching sessions improves patient's knowledge, preparedness and anxiety in relation to chemotherapy | up to 1 month
  To evaluate whether chemotherapy teaching sessions improves patient's knowledge, preparedness and anxiety in relation to chemotherapy
  After informed consent for this study is obtained, patients will be given questionnaire #1 that includes rating their knowledge of the side effects of treatment, their understanding of the treatment schedule, what do in the event of complication, how to reach the medical team and an assessment of the level of anxiety. The questionnaire will be repeated at day 1 of the first chemotherapy treatment to assess the effectiveness of the teaching session. In addition, questionnaire #3 will be administered at day 1 of cycle 2 of their first chemotherapy.

SECONDARY OUTCOMES:
Compare changes in patient's knowledge, preparedness and anxiety in relation to chemotherapy teaching sessions | every 6 months up to two years
  To compare changes in patient's knowledge, preparedness and anxiety in relation to chemotherapy teaching sessions between participating Brown University Oncology Research Group Hospitals After informed consent for this study is obtained, patients will be given questionnaire #1 that includes rating their knowledge of the side effects of treatment, their understanding of the treatment schedule, what do in the event of complication, how to reach the medical team and an assessment of the level of anxiety. The questionnaire will be repeated at day 1 of the first chemotherapy treatment to assess the effectiveness of the teaching session. In addition, questionnaire #3 will be administered at day 1 of cycle 2 of their first chemotherapy.

CONTACTS AND LOCATIONS:
Overall Officials: Anthony Mega, MD, Principal Investigator — Brown University
Locations (4):
- United States (4):
  - Memorial Hospital, Pawtucket, Rhode Island
  - Rhode Island Hospital (including Newport), Providence, Rhode Island
  - The Miriam Hospital, Providence, Rhode Island
  - Roger Williams Medical Center, Providence, Rhode Island